CLINICAL TRIAL: NCT02856178
Title: An Open Label Phase IIa Clinical Study to Evaluate the Safety and Pharmacokinetics of Intravenous and Oral F901318 (Combined With Caspofungin) for Antifungal Prophylaxis in Patients Undergoing Chemotherapy for Acute Myeloid Leukaemia
Brief Title: Study on Safety and Pharmacokinetics of Intravenous F901318 for Fungal Prophylaxis in AML Patients
Acronym: SAFEGUARD
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: study no longer required
Sponsor: F2G Biotech GmbH (Industry)
Collaborators: University Hospital of Cologne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: F901318C20
Record Dates: First submitted 2016-07-14; First posted 2016-08-04 (Estimated); Last update posted 2018-02-15 (Actual); Status verified 2016-08

CONDITIONS: Pulmonary Aspergillosis - Invasive; Acute Myeloid Leukemia
MeSH Terms: conditions — Invasive Pulmonary Aspergillosis; Leukemia, Myeloid, Acute | interventions — olorofim; Caspofungin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- F901318 + Caspofungin (Experimental): Patients will receive F901318 intravenously, starting 24 - 72 h after last chemotherapy infusion:
  * Day 1: 4.0 mg/kg i.v. b.i.d.
  * Day 2 until resolution of neutropenia (max. until day 14): 2.0 mg/kg i.v. b.i.d.
  * Day after last i.v. application: 2.0 mg/kg oral q.d.
  Concomitant medication:
  For Candida prophylaxis, concomitant caspofungin will be administered from the 4th day of chemotherapy until end of neutropenia:
  * Chemo day 4: Caspofungin 70 mg i.v. q.d.
  * Chemo day 5 until resolution of neutropenia or until end of F901318 treatment (day 15): Caspofungin 50 mg i.v. q.d.
  All patients will undergo chemotherapy for acute leukaemia according to local clinical standard.
  Interventions: Drug: F901318; Drug: Caspofungin

INTERVENTIONS:
Drug: F901318 — F901318 treatment starting after completion of chemotherapy. Max. 14 days of intravenous F901318 b.i.d. treatment, followed by one oral dose of F901318. Loading doses 4 mg/kg b.i.d. , maintenance doses 2 mg/kg b.i.d.
Drug: Caspofungin — Intravenous Caspofungin treatment starting during chemotherapy for concomitant prophylaxis of fungal infection. Loading dose 70 mg q.d., maintenance doses 50 mg q.d.
  Other Names: Cancidas®

SUMMARY:
This study assesses the pharmacokinetics and safety of the new antifungal F901318 in AML patients.

DETAILED DESCRIPTION:
F901318 has potent in vitro efficacy against Aspergillus spp. including azole-resistant strains and consistent efficacy in in vivo mouse models of infection. F901318 is active by both oral and intravenous routes of administration in preclinical efficacy studies.

Non-clinical studies and phase I clinical trials show that F901318 has a good overall safety profile and limited potential for drug-drug interactions. F901318 exhibits a highly promising profile which can potentially address the critical treatment requirements for invasive Aspergillus infections in a changing clinical environment in which new classes of antifungals are needed.

This phase IIa study aims to confirm PK and safety information of F901318 from phase I and bridge them to a neutropenic AML patient population, which represents the main population for future efficacy trials. Coadministration of caspofungin will allow recognizing potential factors of suboptimal F901318 exposure without the risk of fatal disseminating infection.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with AML and entering treatment of chemotherapy.
2. Patients are expected to be neutropenic (< 500 ANC/μl) for > 10 days.
3. Provision of written informed consent prior to any study specific procedures.
4. Ability and willingness to comply with the protocol.
5. Patients aged over 18 years.
6. Patient has or will receive within 2 days a multi-lumen central venous catheter as standard of care.

Exclusion Criteria:

1. Documented lung infiltrate at screening.
2. Documented serum GMI ≥0.5 at screening
3. Current IFD or prior history of IFD or patients who received systemic antifungal therapy for proven or probable IFD in the last 12 months.
4. Patients who received any systemic antifungal therapy for more than 72 hours immediately prior to first administration of study medication. Echinocandins and topical polyenes or nystatin are acceptable. Posaconazole and other azoles have to be discontinued at least 3 days before start of F901318.
5. Concomitant exposure to phenobarbital and long acting barbiturates, triazolam, carbamazepine, phenytoin, pimozide, cisapride, efavirenz, ritonavir, rifabutin, rifampicin, ergot alkaloids (ergotamine, dihydroergotamin), ibrutinib, idelalisib, vinca alkaloids, digoxin, dofetilide, quinidine, St. John´s wort, everolimus, sirolimus, astemizole, terfenadine, methadone, alfentanil, fentanyl and other structurally related opiates, warfarin.
6. Documented prolongation of the QTc interval (>450 ms).
7. Concomitant medication that prolongs QT interval (except for cytostatic drugs used during chemotherapy, such as mitoxantrone).
8. Any other concomitant medical condition that, in the opinion of the investigator, may be an unacceptable additional risk to the patient should he/she participate in the study.
9. History of convulsion.
10. Female patients only: Positive result of pregnancy test or breastfeeding.
11. Female patients of childbearing potential who do not agree to not have sexual intercourse during the study or who do not use or do not agree to use appropriate contraceptive methods (prior to and during the study, including 14 days after the last dose of study therapy) as defined in ICH guideline M3(R2) on non-clinical safety studies for the conduct of human clinical trials and marketing authorisation for pharmaceuticals (EMA/CPMP/ICH/286/1995). Hormonal contraception alone is not considered appropriate.
12. Known hypersensitivity to any component of the study medication.
13. A history of additional risk factors for Torsade de pointes (e.g., heart failure, hypokalaemia, cardiomyopathy, sinus bradycardia, symptomatic arrhythmias, family history of long QT Syndrome).
14. Patient has had acute hepatitis in the prior 6 months, chronic hepatitis, cirrhosis (any Child-Pugh class), acute hepatic failure, or acute decompensation of chronic hepatic failure
15. Presence of hepatic disease as indicated by aspartate aminotransferase (AST) or alanine transaminase (ALT)>3 × upper limit of normal (ULN) at Screening. Patients with AST and/or ALT >3 × ULN and <5 × ULN are eligible if these elevations are acute, not accompanied by a total bilirubin ≥2xULN and documented by the investigator as being directly related to an infectious process being treated. During the clinical study, the investigator is responsible for, without delay, determining whether the patient meets potential Hy's law criteria (according to FDA [28]).
16. Patient has a total bilirubin >3 × ULN, unless isolated hyperbilirubinemia is directly related to an acute infection or due to known Gilbert's disease.
17. Calculated creatinine clearance (CrCl) < 50 mL/minute.
18. Medical history of oliguria (< 20 mL/h) unresponsive to fluid challenge.
19. Suspected other or additional cause for neutropenia or immunosuppression (other than AML or myelodysplastic syndrome).
20. Any other medical condition which may affect the clinical evaluability of the patient.
21. Patients previously enrolled in this study.
22. Patient has participated or intends to participate in any other clinical study that involves the administration of an investigational medication at the time of presentation, during the course of the study, or during the 30 days prior to study start. New combinations of labelled substances for chemotherapy are allowed.
23. Chronic ocular disease.
24. Contact lens use intended during study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2017-04-20 (Actual); Study Completion 2017-04-20 (Actual)

PRIMARY OUTCOMES:
Collection of adverse events, results of physical examination, vital signs, ECGs, and laboratory assessments during F901318 intravenous infusion and oral formulation. | 57 days

SECONDARY OUTCOMES:
Concentration-time profile of F901318 following i.v. administration | 14 days
  F901318 trough level assessment for 14 days once per day. On three of these 14 days additional samples for determination of plasma concentration of F901318 will be collected.
Measured concentration of F901318 at the end of an i.v. dosing interval at steady state (Ctrough) | 14 days
Minimum observed plasma or serum, concentration of F901318 during an i.v. dosing interval at steady state (Cmin, ss) | 14 days
Maximum observed plasma or serum, concentration of F901318 during an i.v. dosing interval at steady state (Cmax, ss) | 14 days
Average plasma or serum concentration of F901318 at steady state after i.v. administration (Cav,ss) | 14 days
Area under the concentration-time curve during a F901318 i.v. dosing interval at steady state calculated by trapezoidal rule (AUCT,ss) | 14 days
Area under the concentration vs. time curve from point zero up to the end of infusion of F901318 (AUC(0-T)) | 14 days
  T: total time of infusion
Area under the concentration vs. time curve from time point zero up to the time point t (AUC(0-t)) for F901318 after i.v. administration | 14 days
Area under the concentration vs. time curve from time point zero up to the last measured concentration of F901318 above LOQ (AUC(0-t_last)) after i.v. administration | 14 days
Apparent terminal half-life (t1/2) of F901318 after i.v. administration | 14 days
Terminal rate constant (λz) of F901318 after i.v. administration | 14 days
Apparent clearance (Cl) of F901318 after i.v. administration | 14 days
Plasma concentration of F901318 after oral application | 1 day
  Measurement 2h, 4h, 12h and 24h after oral intake of F901318
Number of patients developing an possible/probable/proven invasive fungal disease (IFD) according to EORTC/MSG criteria | 57 days
  Patients galactomannan index and body temperature will be assessed regularly. If it is clinically indicated the patients will undergo a CT, which will be checked for infiltrations. If infiltrations are detected the patients will undergo a bronchoalveolar lavage, the result of which will be used to analyse BAL GMI, to grow a microbiological culture, to perform histology and perform an Aspergillus PCR. On the basis of the available data for each patient the scientific advisory committee will assess the number of patients suffering from a possible/probable or proven IFD.

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Cornely, PhD, MD, Principal Investigator — University Hospital Cologne

IPD SHARING:
Plan to Share IPD: Undecided